CLINICAL TRIAL: NCT03689335
Title: A Prospective Randomised Controlled Trial of Operative Versus Nonoperative Management of Fractures of the Humeral Diaphysis
Brief Title: HUmeral Shaft Fracture FIXation Study
Acronym: HU-FIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Infirmary of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); University of Edinburgh (Other)
Responsible Party: Principal Investigator, William Oliver, Co-Investigator, Clinical Research Fellow, Royal Infirmary of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/0223
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Closed Fracture of Shaft of Humerus

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial, with 1:1 allocation into one of 2 treatment arms (operative or non-operative treatment). The randomisation is stratified by patient age (<65 years old or ≥65 years old) to ensure approximately equal numbers by age in each treatment arm.
Masking Description: There is no blinding possible in this study, as the presence or absence of a skin incision/surgical scar is obvious to both patient and clinician during follow-up assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Operative (Active Comparator): Surgical fixation of the humeral shaft fracture
  Interventions: Procedure: Operative
- Non-operative (Active Comparator): Conservative treatment of the humeral shaft fracture, using a humeral brace
  Interventions: Device: Humeral brace

INTERVENTIONS:
Procedure: Operative — Open reduction and internal fixation, using a plate and screws (the exact surgical approach and fixation technique utilised will be at the discretion of the treating surgeon)
  Arms: Operative
Device: Humeral brace — Immobilisation in a U-slab or hanging cast, followed by application of a lightweight prefabricated humeral brace
  Arms: Non-operative

SUMMARY:
Fractures of the humeral shaft (upper arm bone) account for approximately 1% of all adult fractures in the United Kingdom. Historically, these injuries have been treated using a cast and/or brace, with immediate surgical fixation reserved for severely- or multiply-injured patients. However, treatment with a brace is associated with several important problems, including poor alignment of the healed bones and shoulder/elbow stiffness. The brace is usually worn for up to 3 months, which interferes with patients' everyday activities and sleeping, and can predispose to skin problems. For 10-15% of patients treated with a brace, their fracture will not heal and will require surgery several months after the original injury, which is more difficult and carries a higher risk of complications. Recent studies suggest that undertaking immediate surgical fixation more often could improve healing and functional outcome for patients with humeral shaft fractures. The only published randomised controlled trial (RCT) to date showed no difference in clinical outcome between conservative and operative management; unfortunately, however, the operative technique used was unusual and would be considered highly suboptimal in most Western countries.

This study will include adult patients (≥16 years), with capacity to consent and complete post-operative questionnaires in English, presenting to a single Orthopaedic trauma unit. Participants will be randomised to either non-operative treatment (with a brace) or operative treatment (i.e. surgical fixation). The investigators will assess whether there is a difference between the groups in terms of patient-reported outcome scores, fracture healing, complications, pain and return to work/sport over a one-year follow-up period. Participants will be enrolled into the study after obtaining informed consent. Following randomisation (to either non-operative treatment or surgical fixation), participants will then be reviewed at several defined timepoints, with a combination of clinical examination, X-rays and patient-reported outcome scores. The investigators hope that study results will enable surgeons to make better-informed decisions when managing patients with humeral shaft fractures.

DETAILED DESCRIPTION:
This study will include patients presenting to a single centre - the Edinburgh Orthopaedic Trauma Unit, Royal Infirmary of Edinburgh - with an isolated fracture of the humeral shaft.

All patients will be treated in the Emergency Department (ED) with closed reduction and application of a U-slab or hanging cast, and then referred to the Orthopaedic service. This referral will occur just prior to discharge from the ED, and will either be immediate (via the on-call team, for example where the patient requires in-patient admission) or delayed (via the Trauma Triage Clinic system, in which patients are discharged home and subsequently given an outpatient appointment).

Patients will be considered for the study if the following initial criteria are met:

1. The patient has sustained a fracture of the humeral shaft (defined as any fracture in which the major fracture line does not extend to within one metaphyseal width/'Müller box' of either the shoulder or elbow joint);
2. The patient is aged 16 years or older;
3. The patient is able to comply with post-operative data gathering, including attending local follow-up appointments and completing questionnaires in English.

Complete inclusion and exclusion criteria are provided in the 'Eligibility' section.

All adult patients presenting with a humeral shaft fracture that satisfy the inclusion criteria will be invited to participate in the study. Patients are eligible for enrolment in the study regardless of sex, race or ethnicity. Vulnerable populations, including patients unable to give informed consent and complete post-operative questionnaires in English, will not be recruited.

Patients will be predominately recruited either in the ED, on the Orthopaedic ward (if they are admitted), or at the first outpatient clinic appointment (approximately 1-2 weeks following their injury). The treating clinical team will introduce appropriate patients to the study and initiate the process of informed consent. A patient information sheet will be provided for them to read before agreeing to take part.

Whether potential participants are identified and introduced to the study in the ED, on the Orthopaedic ward, or in the outpatient clinic (which the investigators anticipate to be the most common scenario), they will have until 2 weeks post-injury to decide whether or not to take part. For practical reasons, performing surgery on a humeral shaft fracture that is older than 3 weeks is more challenging (as the healing process has already begun), and therefore the investigators ask any potential participants to make their decision by the 2-week mark so that surgery can be scheduled (if appropriate).

If the patient agrees, a member of the research team will review the study protocol in detail and address any questions the patient may have. If the patient is willing to participate, the research team member will complete the informed consent process. If this is during an out-of-hours period, consent will be taken by the appropriately qualified on-call Orthopaedic trainee or consultant. All trainees and consultants within the Unit will have ongoing briefing regarding the aims and methodology of the study. With the permission of the patient, a letter will be sent to their General Practitioner informing them of their involvement in the study.

Patients will be given a copy of their consent form, and informed that their participation is voluntary and that they can withdraw at any time during the study without any detriment to their normal care. Patients may take as long as they like to consider participation, provided they still meet all the inclusion criteria (below) and surgery (if appropriate) can be performed within 3 weeks of injury. Patients requiring a longer period of time consider their participation than is feasible at the first meeting will be contacted the following day for a further discussion, either face-to-face or over the telephone. They will also be given the contact details of an Orthopaedic specialist independent of the study, to allow them access to further information if they so require.

Upon agreeing to take part, patients will be randomised to either operative or non-operative management of their humeral shaft fracture. On enrolment, a data collection form will be started with demographic and injury-related information collected. Regardless of the treatment arm, patients will be followed-up in person at the following post-intervention stages: 2 weeks, 6 weeks, 12 weeks, 26 weeks and 52 weeks.

Patients randomised to operative management of their humeral shaft fracture will undergo surgical fixation using a standard technique of plating and screw fixation. The exact surgical approach and fixation technique utilised will be at the discretion of the treating surgeon. Similarly, post-operative immobilisation and range-of-motion restrictions will be at the discretion of the treating surgeon. This is determined by a number of factors including the injury/fracture pattern, bone quality, co-morbidities and patient compliance.

Patients randomised to non-operative management will be managed as per current standard practice for our Unit. This involves a period of immobilisation in a U-slab or hanging cast for up to 2 weeks, before application of a lightweight prefabricated humeral brace in the outpatient clinic. Patients will be permitted to start passive pendular shoulder exercises with full elbow, wrist and hand mobilisation as soon as the humeral brace has been applied. Post-operative physiotherapy will be arranged at the discretion of the treating surgeon, as occurs in everyday clinical practice.

The primary outcome measure is the Disabilities of the Arm, Shoulder and Hand (DASH) score at 3 months post-intervention. Prior to study commencement, a prospective power calculation was used to determine the number of patients required in each treatment group. The minimal clinically-important difference in the DASH score is reported to be 10 points, and the assumed standard deviation is 12 points for both the operative and non-operative groups. Thus, using a 2-sided t-test with a 5% significance, a total of 70 patients (35 in each group) are required to produce a 90% power to detect a meaningful difference in the DASH score at 3 months between the 2 groups, assuming a 10% loss-to-follow-up. Statistical analysis for the study will be performed by an independent statistician, employed through the local University Statistics department.

Further details regarding the primary outcome measure and secondary outcome measures are provided in the 'Outcome Measures' section.

All follow-up assessment will take place during outpatient clinic visits, initially with the treating consultant surgeon's team. Follow-up assessment will be undertaken over a one-year period (2 weeks, 6 weeks, 12 weeks, 26 weeks and 52 weeks). Routine follow-up in our institution for patients with a humeral shaft fracture is outpatient review with radiographs at 2 weeks, 6 weeks and 12 weeks, although additional follow-up is sometimes required if there are problems with ongoing pain or inadequate fracture healing. At most, therefore, study participants will attend 2 additional clinic appointments compared to patients treated outwith the study.

At each clinic visit, the treatment group (i.e. operative or non-operative) will be specified, a physical examination will be performed, and treatment complications and the need for re-operation will be recorded. Patients will be given time to complete a self-reported questionnaire, which will generate clinical outcome scores.

The investigators will also review electronic patient records, to assess whether any patient underwent subsequent surgery on the affected arm during the study period. This would include debridement/irrigation for infection and/or removal of metalwork.

ELIGIBILITY:
Inclusion Criteria:

1. Fracture of the humeral shaft
2. Closed injury
3. Age ≥16 years
4. Able to provide informed consent in English
5. Surgery performed within 3 weeks of date of injury

Exclusion Criteria:

1. Completely undisplaced fractures
2. Injuries considered to be an absolute indication for surgery (including severe associated neurovascular injury, open fractures and bilateral injuries)
3. Patients with a periprosthetic or pathological fracture
4. Patients with an additional spine or limb injury (including those with polytrauma), which may impact upon functional rehabilitation
5. Patients medically unfit for surgery
6. Very frail patients (CSHA Clinical Frailty Score ≥6/9)
7. Pregnant women with predetermined treatment
8. Patients declining operative management
9. Patients unable to provide informed consent in English
10. Patients unable to comply with post-operative data gathering, including completing questionnaires in English
11. Non-residents, unable to return to the Unit for follow-up for a period of 1-year
12. Where the treating surgeon does not feel that inclusion in the trial is in the patient's best interests, either due to fracture pattern or patient factors

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) score | 3 months
  The DASH score is a functional rating scale developed in 1996, which has been used extensively as a research tool in upper limb surgery. It consists of a 30-item self-reported questionnaire, and 2 optional modules assessing work and sports/performing arts. Patient symptoms (including pain, weakness, stiffness and tingling/numbness) and functional status (including physical, social and psychological aspects) during the week prior to survey completion are assessed. A final score is awarded from 0 to 100, with 0 representing no disability and 100 the worst possible disability. The DASH score at 3 months post-intervention will form the primary outcome measure.

SECONDARY OUTCOMES:
Change in Disabilities of the Arm, Shoulder and Hand (DASH) score | 6 weeks, 3 months, 6 months, one year
  The DASH score is a functional rating scale developed in 1996, which has been used extensively as a research tool in upper limb surgery. It consists of a 30-item self-reported questionnaire, and 2 optional modules assessing work and sports/performing arts. Patient symptoms (including pain, weakness, stiffness and tingling/numbness) and functional status (including physical, social and psychological aspects) during the week prior to survey completion are assessed. A final score is awarded from 0 to 100, with 0 representing no disability and 100 the worst possible disability. Change in the DASH score over the one-year follow-up period will form a secondary outcome measure.
Pain visual analogue scale (VAS) | 2 weeks, 6 weeks, 3 months, 6 months, one year
  Assessment of pain in the injured arm, from 0 (no pain) to 10 (worst pain imaginable).
Treatment complications | 2 weeks, 6 weeks, 3 months, 6 months, one year
  Complications of treatment, including neurovascular injury, superficial/deep infection, failure of fixation, revision surgery, skin complications (including eczema and cellulitis) and complex regional pain syndrome (CRPS).
Return to work/sport | 6 weeks, 3 months, 6 months, one year
  Time taken to return to work and sport (if relevant).
Satisfaction with service visual analogue scale (VAS) | 2 weeks, 6 weeks, 3 months, 6 months, one year
  Assessment of overall satisfaction with clinical care provided, from 0 (completely dissatisfied) to 100 (completely satisfied).
Shoulder/elbow range of motion (measured in degrees) | 6 weeks, 3 months, 6 months, one year
  Recovery of shoulder and elbow range of motion over the one-year follow-up period. This will be assessed through clinical measurement of shoulder elevation, abduction, external and internal rotation, and elbow flexion and extension.
Radiographic assessment | 6 weeks, 3 months, one year
  Standard anteroposterior and lateral X-rays of the humerus over the one-year follow-up period. These X-rays will be used to assess progression of fracture healing, as well as the final humeral deformity (measured in degrees) in the coronal (varus/valgus) and sagittal (procurvatum/recurvatum) planes once healing has occurred.
EuroQol (EQ-5D) Health Outcome score | 6 weeks, 3 months, 6 months, one year
  A standardised instrument for use as a measure of health outcome.
12-item Short Form (SF-12) Health Survey score | 6 weeks, 3 months, 6 months, one year
  A standardised instrument for use as a measure of health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel G Molyneux, FRCSEd (Tr&Orth), Principal Investigator — Royal Infirmary of Edinburgh
Locations (1):
- Edinburgh Orthopaedic Trauma Unit, Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oliver WM, Carter TH, Graham C, White TO, Clement ND, Duckworth AD, Molyneux SG. A prospective randomised controlled trial of operative versus non-operative management of fractures of the humeral diaphysis: the HUmeral Shaft Fracture FIXation (HU-FIX) Study protocol. Trials. 2019 Aug 5;20(1):475. doi: 10.1186/s13063-019-3576-0. PMID 31383027
- [Derived] Oliver WM, Bell KR, Carter TH, Graham C, White TO, Clement ND, Duckworth AD, Molyneux SG. Operative vs Nonoperative Management of Fractures of the Humeral Diaphysis: The Humeral Shaft Fracture Fixation Randomized Clinical Trial. JAMA Surg. 2025 May 1;160(5):508-516. doi: 10.1001/jamasurg.2025.0301. PMID 40136271